CLINICAL TRIAL: NCT02930083
Title: Validating Three Common Occupational Therapy Assessments in Participants With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, LEE SHU CHUN, Occupational Therapist, Taipei City Hospital
Other Study IDs: OT-3tools-2014
Record Dates: First submitted 2016-10-09; First posted 2016-10-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
To improve activities of daily living (ADL) and social functions is the important treatment plans and goals in participants with schizophrenia. Precise and effective measures of ADL and social functions are critical for clinicians to set up appropriate treatments plans, follow up participants' changes, and understand participants' progress. Three common measures of ADL and social functions used in participants with schizophrenia were the Comprehensive Occupational Therapy Evaluation Scale (COTES), the Activities of Daily Living Rating Scale third ed. (ADLRS-3), and the Social Functioning Scale. To investigators' knowledge, psychometric properties of these assessments have not been examined in participants with schizophrenia. Therefore, the purpose of the study is to (1) examine internal consistency and construct validity of these 3 assessments (the COTES, the ADLRS-3, and the Social Functioning Scale); and (2) calculate missing rate of self-report assessment (the ADLRS-3 and the Social Functioning Scale). Investigators expect that these results of internal consistency, construct validity and/or missing rate will provide empirical evidence for using these three measures in both clinical and research setting.

DETAILED DESCRIPTION:
Social dysfunction is one of the main characteristics of participants with schizophrenia and influences participants' daily functions and quality of life. The Social Functioning Scale-Taiwan short form (SFST) is commonly used to measure social function in participants with schizophrenia. However, no study has examined psychometric properties of the SFST in participants with schizophrenia exclusively. Therefore, the study aimed to examine missing rate, ceiling effect/floor effect, internal consistency, and convergent validity of the SFST in participants with schizophrenia. Investigators obtained schizophrenic self-report data (the SFST and the ADLRS-3) from occupational therapy records. The Chinese version of the Activities of Daily Living Rating Scale (ADLRS-3), which has 10 domains, is commonly used for assessing activities of daily living (ADL) in participants with schizophrenia. However, construct validity (i.e., unidimensionality) for each domain of the ADLRS-3 is unknown, limiting the explanations of the test results. From occupational therapy records, investigators obtained self-report data of the ADLRS-3. Confirmatory factor analysis (CFA) was conducted to examine the 10 one-factor structures. If a domain showed an insufficient model fit, exploratory factor analysis (EFA) was performed to investigate the factor structure and choose one factor representing the original construct. Internal consistency was examined using Cronbach's alpha. Ceiling and floor effects were determined by the percentage of participants with the maximum and minimum scores in each domain, respectively. To evaluate construct validity (i.e., unidimensionality and convergent validity) and Rasch reliability of the Comprehensive Occupational Therapy Evaluation Scale (COTES) in participants with schizophrenia. From occupational therapy records, investigators collected COTES data of participants with schizophrenia. The 20-item COTES contains three subscales. For construct validity, investigators first examined the unidimensionality of each subscale using Rasch analysis. After unidimensionality was supported, investigators examined convergent validity using Pearson's r and Rasch reliability of the individual subscales in unidimensional and multidimensional approaches.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with schizophrenia

Exclusion Criteria:

* participants who had a history of severe brain injury
* diagnoses of mental retardation or substance abuse

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective study was conducted and the data were obtained from occupational therapy records at community rehabilitation centers in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Social Functioning Scale-Taiwan short form Social Functioning Scale-Taiwan short form | Sep. 2012 to Dec. 2014
Activities of Daily Living Rating Scale III | Sep. 2012 to Dec. 2014
Comprehensive Occupational Therapy Evaluation Scale | Sep. 2012 to Dec. 2014